CLINICAL TRIAL: NCT03944785
Title: A Prospective, Observational Study to Evaluate Changes in Non-Motor Symptoms and Other Clinical Outcome Assessments of Parkinson's Disease Patients Treated With XADAGO (Safinamide)Tablets
Brief Title: Clinical Outcome Assessment of Parkinson's Disease Patients Treated With XADAGO (Safinamide)
Acronym: PRO-Go
Status: Completed | Type: Observational
Sponsor: Supernus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: USWM-SA1-4001
Record Dates: First submitted 2019-05-01; First posted 2019-05-10 (Actual); Results first posted 2021-02-18 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2021-07

CONDITIONS: Idiopathic Parkinson Disease
Keywords: Parkinson's disease; Safinamide; Xadago; MAO-B inhibitor; off; non-motor symptoms; motor symptoms; levodopa; PD
MeSH Terms: conditions — Parkinson Disease | interventions — safinamide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Parkinson's Disease Patients: PD patients who have been newly prescribed safinamide (XADAGO) for the treatment of OFF episodes as described in the XADAGO Package Insert
  Interventions: Drug: XADAGO (safinamide)

INTERVENTIONS:
Drug: XADAGO (safinamide) — XADAGO (safinamide) is a monoamine oxidase type B (MAO-B) inhibitor indicated as adjunctive treatment to levodopa/carbidopa in patients with Parkinson's disease experiencing off episodes.
  Other Names: XADAGO; safinamide

SUMMARY:
This is a Phase IV, prospective, observational, post-marketing study designed to obtain additional data on the effect of XADAGO on motor and non-motor symptoms in Parkinson's Disease patients newly prescribed XADAGO.

DETAILED DESCRIPTION:
This Phase IV, multicenter, prospective, observational study to evaluate clinician-reported outcomes and patient-reported outcomes related to motor and non-motor symptoms, health status, quality of life and treatment satisfaction in PD patients who have been newly prescribed XADAGO according to Package Insert indication.

This study also will gather "real world" data from a PD population in the US regarding their overall experience and degree of satisfaction with the use of XADAGO as an add-on treatment to their L-dopa regimen. Treatment experience will be captured using patient self-rating assessments as well as clinician ratings on assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Patient (and Care Partner, if required per Inclusion Criterion 6) is able to understand and provide signed informed consent and HIPAA authorization in English.
2. Patient with diagnosis of idiopathic PD (all stages).
3. Independent of the study, clinician's and patient's choice of treatment is XADAGO in accordance with the Package Insert indication.
4. Patient is willing and able to participate in the study and complete study-related assessments for 2 months and, patients can continue for an optional 4-month study extension.
5. Patient has access to an electronic device for the interim completion of PROs.
6. Patient has an available Care Partner who is able and willing to assist with clinic attendance and completion of study assessments (e.g., PROs, health outcomes, etc.), if in the PI's opinion, assistance is needed to comply with all study visits and procedures.

Exclusion Criteria:

1. Any of the warnings, precautions, or contraindications listed in the XADAGO Package Insert that in the opinion of the PI would prevent appropriate treatment with XADAGO or impair study participation (e.g., pregnancy, lactation, severe hepatic impairment, etc.).
2. Participation in any other clinical trial of an investigational drug or device within 4 weeks prior to the Baseline Visit or at any time during the study.
3. Patient is currently receiving chemotherapy or radiation for any form of cancer (if history of cancer, must be in clinical remission at study entry) or currently receiving immunotherapy.
4. Patients with conditions that are likely to prevent them from accurately and reliably completing study assessments, including evidence of moderate or severe dementia as determined by the clinician (not to include mild cognitive impairment [MCI]); major psychiatric illness (specifically diagnosis of schizophrenia, bipolar disorder or a history of attempted suicide); and/or severe and progressive medical illness (including terminal cancer, end-stage renal disease +/- undergoing dialysis).
5. Severe or unpredictable dyskinesia at the time of the Baseline Visit.
6. Previous participation in this study; a patient may not re-enroll after prior discontinuation or completion

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Parkinson's Disease patients who have been newly prescribed XADAGO
Sampling Method: Non-Probability Sample
Enrollment: 164 (Actual)
Dates: Start 2017-11-30 (Actual); Primary Completion 2019-12-23 (Actual); Study Completion 2020-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Najeebah Abdul-Musawir, MD,MBA, Study Director — Supernus Pharmaceuticals, Inc.
Locations (30):
- United States (30):
  - Alabama Neurology Associates, Homewood, Alabama
  - Movement Disorders Neurology, Inc., Bakersfield, California
  - B.E.S.T. Center of Orange County, Laguna Hills, California
  - Valley Parkinson Clinic, Los Gatos, California
  - UC Davis Medical Center, Sacramento, California
  - Hartford Healthcare, Vernon, Connecticut
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - Parkinson's Disease and Movement Disorders Center of Boca Raton, Boca Raton, Florida
  - Neuron Research, Naples, Florida
  - Parkinson's Disease Treatment Center of SW Florida, Port Charlotte, Florida
  - Sarasota Memorial Hospital Clinical Research Cener, Sarasota, Florida
  - Central DuPage Hospital, Winfield, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Baptist Health System, Richmond, Kentucky
  - Southeast Neuroscience Center, LLC, Gray, Louisiana
  - Lester and Cox Medical Center, Springfield, Missouri
  - Neurological Associates of Long Island, PC, Lake Success, New York
  - NYU Winthrop Hospital, Mineola, New York
  - FryeCare Neurology, Hickory, North Carolina
  - Dayton Center for Neurological Disorders, Centerville, Ohio
  - The Movement Disorder Clinic of Oklahoma, Tulsa, Oklahoma
  - Neurology and Stroke Associates, Lititz, Pennsylvania
  - Prisma Health, Greenville, South Carolina
  - Covenant Medical Group, Lubbock, Texas
  - Texas Institute for Neurological Disorders, Sherman, Texas
  - Houston Methodist - Sugar Land, Sugar Land, Texas
  - Baylor Scott and White Health, Temple, Texas
  - Inova Medical Group- Neurology I, Alexandria, Virginia
  - Meridian Clinical Research, LLC, Norfolk, Virginia
  - Puget Sound Neurology, Tacoma, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- DA Switchers: Parkinson's Disease patients that have switched to safinamide (XADAGO) from a dopamine agonist (DA)
- MAO-B Switchers: Parkinson's Disease patients that have switched to safinamide (XADAGO) from a monoamine oxidase-B (MAO-B) inhibitor
- MAO-B Naive: Parkinson's Disease patients taking safinamide (XADAGO) that are MAO-B inhibitor naïve.
Period: 2 Month Study Completion
Arm/Group | DA Switchers | MAO-B Switchers | MAO-B Naive
Started (Participants were prospectively followed for 2 months.) | 2 | 34 | 128
Completed | 2 | 30 | 123
Not Completed | 0 | 4 | 5
Period: 4 Month Study Optional Extension
Arm/Group | DA Switchers | MAO-B Switchers | MAO-B Naive
Started (Continued participation for 4 additional months as an optional extension to the original 2 months.) | 1 | 10 | 64
Completed | 0 | 8 | 41
Not Completed | 1 | 2 | 23

BASELINE CHARACTERISTICS:
Population: Safety Population: All patients who sign informed consent for the study, complete baseline assessments, and receive at least 1 dose of XADAGO.
Groups:
- MAO-B: Parkinson's Disease patients that have switched to safinamide (XADAGO) from a monoamine oxidase-B (MAO-B) inhibitor
- Total: Total of all reporting groups
Arm/Group | DA Switchers | MAO-B | MAO-B Naive | Total
Number analyzed (Participants) | 2 | 34 | 128 | 164
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.5 (6.36) | 65.3 (8.28) | 68.1 (7.77) | 67.4 (7.92)
Age, Customized [Count of Participants; unit: Participants]
  Age 30-65 | 1 | 16 | 39 | 56
  Age >= 65 | 1 | 18 | 89 | 108
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 6 | 43 | 49
  Male | 2 | 28 | 85 | 115
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 6 | 6
  Not Hispanic or Latino | 2 | 34 | 122 | 158
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 3 | 4 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 1 | 2
  White | 2 | 30 | 121 | 153
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 2 | 2
Height (cm) [Mean (Standard Deviation); unit: cm] | 179.6 (6.51) | 173.1 (11.67) | 171.0 (11.91) | 171.6 (11.83)
Weight (kg) [Mean (Standard Deviation); unit: kg] | 96.2 (0.64) | 85.0 (16.95) | 88.1 (22.60) | 87.6 (21.42)
BMI (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 29.9 (2.36) | 28.4 (5.17) | 30.1 (7.05) | 29.7 (6.68)
Movement Disorders Society - Unified Parkinson's Disease Rating Scale [Mean (Standard Deviation); unit: units on a scale] — MDS-UPDRS: 4-part assessment of the multiple clinical disabilities of Parkinson's Disease. Part I (13 items; Score 0-52) examines non-motor experiences, Part II (13 items; Score 0-52) examines motor experiences, Part III (33 items; Score 0-132) examines the cardinal motor disabilities and Part IV (6 items; Score 0-24) examines motor complications. Each Part has 0-4 ratings, where 0 (no problems) to 4 (severe problems) and scores for each part are summed to calculate the total score which ranges from 0-260. Higher scores represent worse outcomes for each part and total score. Population: Evaluable Population: All patients in the safety population who complete at least the Movement Disorders Society - Unified Parkinson's Disease Rating Scale assessment at the Study Day 60 visit
  units on a scale
    Part 1: number analyzed (Participants) | 2 | 28 | 123 | 153
    Part 1 | 12.0 (2.83) | 10.5 (6.32) | 12.3 (6.88) | 11.9 (6.75)
    Part 2: number analyzed (Participants) | 2 | 28 | 123 | 153
    Part 2 | 7.0 (4.24) | 11.8 (9.21) | 13.8 (8.66) | 13.3 (8.75)
    Part 3: number analyzed (Participants) | 2 | 28 | 123 | 153
    Part 3 | 24.0 (2.83) | 23.4 (14.13) | 30.0 (26.0) | 28.7 (15.95)
    Part 4: number analyzed (Participants) | 2 | 28 | 123 | 153
    Part 4 | 3.0 (0.00) | 5.3 (3.81) | 4.5 (4.04) | 4.6 (3.98)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Movement Disorders Society -Unified Parkinson's Disease Rating Scale (MDS-UPDRS)
Description: MDS-UPDRS: 4-part assessment of the multiple clinical disabilities of Parkinson's Disease. Part I (13 items; Score 0-52) examines non-motor experiences, Part II (13 items; Score 0-52) examines motor experiences, Part III (33 items; Score 0-132) examines the cardinal motor disabilities and Part IV (6 items; Score 0-24) examines motor complications. Each Part has 0-4 ratings, where 0 (no problems) to 4 (severe problems) and scores for each part are summed to calculate the total score which ranges from 0-260. Higher scores represent worse outcomes for each part and total score.
Time Frame: Baseline to Study Day 60
Population: Overall Number of Participants Analyzed represented by initial number analyzed at study visit Day 60; Number may differ for each Part (1-4) due to availability of score data. Evaluable Population: all subjects in the safety population who complete at least the MDS-UPDRS assessment at the Study Day 60 visit. Evaluable population will be used to analyze MDS-UPDRS endpoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DA Switchers | MAO-B Switchers | MAO-B Naive
Number analyzed (Participants) | 2 | 28 | 120
score on a scale
  Part 1 | -5.0 (5.66) | -1.0 (5.13) | -1.9 (6.16)
  Part 2 | 0.0 (2.83) | -2.3 (5.40) | -2.6 (5.28)
  Part 3: number analyzed (Participants) | 2 | 28 | 115
  Part 3 | 1.5 (2.12) | -3.3 (7.78) | -4.5 (11.10)
  Part 4: number analyzed (Participants) | 2 | 28 | 119
  Part 4 | -0.5 (3.54) | -0.3 (3.28) | -0.2 (3.05)

2. Primary Outcome: Change From Baseline in Parkinson's Disease Questionnaire (PDQ-39) Scores
Description: PDQ-39 is a patient-reported outcome designed to address aspects of functioning and well-being for those affected by PD. Each of the 39 items is rated using a 5 point Likert scale with 0 for never having difficulties/problems and 4 for always having difficulties/problems. The sum score of the 39 items will be calculated and used for analysis, with scores ranging from 0-156. Higher scores indicate worse outcomes.
Time Frame: Baseline to Study Day 60
Population: Overall Number of Participants Analyzed represented by number analyzed at study visit Day 60. Safety Population: all subjects who sign informed consent form, complete baseline assessments, receive at least 1 dose of XADAGO. Safety population used to analyze all efficacy endpoints except MDS-UPDRS.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DA Switchers | MAO-B Switchers | MAO-B Naive
Number analyzed (Participants) | 1 | 25 | 97
score on a scale | -1.8 | 0.5 (9.73) | -0.5 (9.90)

3. Primary Outcome: Change From Baseline in Montreal Cognitive Assessment (MoCA) Total Score.
Description: MoCA is a 30-point, 1-page test designed to assess several cognitive domains, including visuospatial abilities (5 points), naming (3 points), attention (6 points), language (3 points), abstraction (2 points), delayed recall (5 points), and orientation to time and place (6 points). The total score ranges from 0 to 30, with higher scores indicating better performances.
Time Frame: Baseline to Study Day 60
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DA Switchers | MAO-B Switchers | MAO-B Naive
Number analyzed (Participants) | 2 | 28 | 119
score on a scale | 0.0 (1.41) | 0.9 (2.41) | 0.4 (2.45)

4. Primary Outcome: Treatment Satisfaction Questionnaire for Medication (TSQM-9) Scores
Description: TSQM-9 consists of 9 questions to assess patients' satisfaction with medication using a range of responses from 1 (extremely dissatisfied) to (7 extremely satisfied). This patient reported outcome provides scores on three parts: effectiveness, convenience, and global satisfaction. The sum of the 9-questions will be calculated and used for analysis. The total score ranges from 0 to 63, with higher scores indicating better treatment satisfaction.
Time Frame: Study Day 60
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DA Switchers | MAO-B Switchers | MAO-B Naive
Number analyzed (Participants) | 1 | 25 | 99
score on a scale | 56.0 | 38.9 (7.73) | 41.0 (9.81)

5. Primary Outcome: Clinical Global Impression of Change (CGI-C)
Description: CGI-C is a 7-point scale depicting a Principal Investigator or certified Health Care Professional designee rating of the patient's overall improvement using a range of responses from a minimum of 1 (very much improved) to a maximum of 7 (very much worse).
Time Frame: Study Day 60
Measure: Count of Participants; unit: Participants
Arm/Group | DA Switchers | MAO-B Switchers | MAO-B Naive
Number analyzed (Participants) | 2 | 34 | 128
Participants
  Very Much Improved | 0 | 1 | 13
  Much Improved | 1 | 7 | 29
  Minimally Improved | 0 | 10 | 38
  No Change | 1 | 6 | 31
  Minimally Worse | 0 | 2 | 7
  Much Worse | 0 | 1 | 3
  Very Much Worse | 0 | 0 | 0

6. Primary Outcome: Patient Global Impression of Change (PGI-C)
Description: PGI-C is a 7-point scale depicting a patient's rating of overall improvement using a range of responses from 1 (very much improved) to 7 (very much worse).
Time Frame: Study Day 60
Population: Participants Analyzed does not match the Participant Flow because some patient data was not captured for the visit. Safety Population: all subjects who sign informed consent form, complete baseline assessments, receive at least 1 dose of XADAGO. Safety population used to analyze all efficacy endpoints except MDS-UPDRS.
Measure: Count of Participants; unit: Participants
Arm/Group | DA Switchers | MAO-B Switchers | MAO-B Naive
Number analyzed (Participants) | 2 | 25 | 100
Participants
  Very Much Improved | 0 | 1 | 9
  Much Improved | 2 | 3 | 25
  Minimally Improved | 0 | 9 | 31
  No Change | 0 | 8 | 30
  Minimally Worse | 0 | 2 | 2
  Much Worse | 0 | 2 | 2
  Very Much Worse | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | DA Switchers | MAO-B Switchers | MAO-B Naive
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/34 | 2/128
Serious Adverse Events (participants affected / at risk) | 0/2 | 2/34 | 8/128
Other Adverse Events (participants affected / at risk) | 1/2 | 8/34 | 17/128
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DA Switchers (N=2) | MAO-B Switchers (N=34) | MAO-B Naive (N=128)
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Postoperataive ileus (Gastrointestinal disorders) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1
Traumatic haemothorax (Injury, poisoning and procedural complications) | 0 | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Dysarthria (Nervous system disorders) | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DA Switchers (N=2) | MAO-B Switchers (N=34) | MAO-B Naive (N=128)
Nausea (Gastrointestinal disorders) | 0 | 3 | 9
Dizziness (Nervous system disorders) | 0 | 2 | 4
Tremor (Nervous system disorders) | 1 | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 2 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-10-12): https://cdn.clinicaltrials.gov/large-docs/85/NCT03944785/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-08): https://cdn.clinicaltrials.gov/large-docs/85/NCT03944785/SAP_001.pdf